CLINICAL TRIAL: NCT06362902
Title: Laparoscopic Right Hemicolectomy With Transrectal Specimen Extraction for Colon Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Haitao Zhou, Clinical Professor, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOSES-VIII B
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Colon Cancer
Keywords: Colon cancer; Laparoscopic Right Hemicolectomy; Natural orifice specimen extraction surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Right Hemicolectomy With Transrectal Specimen Extraction (Experimental): STEP 1: Dissection and separation The mesentery and vessels were dissected and separated according to the principle of complete mesocolic excision.
  STEP 2: Intracorporeal anastomosis An enterotomy was performed on the antimesenteric side of the ileum at the edge of the staple line. This maneuver was replicated on the transverse colic side. Subsequently, the cartridge jaw of the stapler was inserted into the transverse colon. The stapler was fired and withdrawn, and the common enterotomy was sealed by using another linear stapler.
  STEP 3: Transrectal specimen extraction A longitudinal incision was made on the anterior of wall of the upper rectum. The assistant employed oval forceps to extract the specimen along with the protective sleeve through the incision in the upper rectum. After the complete extraction of the specimen, a full-layer running suturing was performed to close the incision.
  Interventions: Procedure: Laparoscopic right hemicolectomy with transrectal specimen extraction

INTERVENTIONS:
Procedure: Laparoscopic right hemicolectomy with transrectal specimen extraction — Laparoscopic right hemicolectomy with transrectal specimen extraction

SUMMARY:
The purpose of this study is to investigate the preliminary surgical outcomes of laparoscopic right hemicolectomy with transrectal specimen extraction. The hypothesis is that this type of natural orifice specimen extraction surgery (NOSES) could achieve good short-term and oncological outcomes for right colon cancer patients.

DETAILED DESCRIPTION:
This study is a prospective single-arm clinical study. 37 patients with right colon cancer undergoing laparoscopic right hemicolectomy with transrectal specimen extraction are planned to be included in the study. The purpose of this study is to investigate the preliminary surgical outcomes of laparoscopic right hemicolectomy with transrectal specimen extraction. The primary endpoint is the postoperative complications of this type of natural orifice specimen extraction surgery (NOSES). The primary hypothesis is that NOSES could reduce postoperative complications. In addition, operating time, intraoperative bleeding, post-operative recovery and quality of life (QoL) are secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven colon carcinoma;
2. Imaging diagnosis of T1-3 colon cancer;
3. The tumor located in the cecum, ascending colon, or colonic hepatic flexure;
4. Maximal tumor diameter ≤5 cm;
5. Body mass index (BMI) ≤30 kg/m2;
6. Written informed consent;

Exclusion Criteria:

1. Complete intestinal obstruction;
2. Hepatitis activity and peripheral neuropathy (such as peripheral neuritis, pseudo meningitis, motor neuritis, and sensory impairment);
3. Significant organ dysfunction or other significant diseases, including clinically relevant coronary artery disease, cardiovascular disease, or myocardial infarction within the 12 months before enrollment; severe neurological or psychiatric history; severe infection; active disseminated intravascular coagulation;
4. Pregnancy or breastfeeding;
5. Alcohol abuse or drug addiction;
6. Concurrent uncontrolled medical condition;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The rate of postoperative complications | up to 30 days
  The rate of postoperative complications = patients with any postoperative complications/all cases.

SECONDARY OUTCOMES:
Operating time | up to 1 days
  Operating time = The Operative time was defined as the time first skin incision was made to final skin closure
Estimated blood loss | up to 1 days
  Estimated blood loss = The sum of the blood in the suction canister (the total volume after subtracting the amount of irrigation fluid used) and the segment of increased weight of swabs used during operation phase (1 ml of blood is about weighs 1g)
The time of first flatus | up to 5 days
  The time of first flatus = The time of first flatus reported by patients
Postoperative hospitalization | up to 30 days
  Postoperative hospitalization = the number of nights from surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Zhou, M.D., Study Chair — National Cancer Center, China
Locations (1):
- National Cancer Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Participants' data are only allowed to be used for the analysis of this study and are not authorized to be shared with other researchers.